CLINICAL TRIAL: NCT03444233
Title: Impact of Short-term Fructose-enriched Diet on Serum Metabolome by Normal- and Over-weighed Women.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Fructose Study
Record Dates: First submitted 2018-02-16; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Diet

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low f1 diet (Experimental): low fructose diet week 1
  Interventions: Other: Diet
- fruit rich diet (Experimental): fruit rich diet week 2
  Interventions: Other: Diet
- low f2 diet (Experimental): low fructose diet week 3
  Interventions: Other: Diet
- HFCS rich diet (Experimental): HFCS rich diet week 4
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — 7 days fruit-rich diet, 7 days HFCS-rich diet
  Other Names: C-TruSweet 01750, Cargill Deutschland GmbH, Krefeld

SUMMARY:
The purpose of this study is to investigate how a high-fructose diet, either by high fructose intake from complex, natural foods or by fortifying the diet with corn syrup, affects the metabolism. Furthermore, it will be investigate if there are differences between obese and normal weight participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, aged between 20 and 30 years
* normal weighted (BMI ≤ 25 kg/m2) and obese (BMI 35-50 kg/m2)
* written informed consent

At initial medical examination an anamnesis, physical examination, blood sample collection (10 ml) was performed to check for eligibility. Furthermore, a hydrogen breath test was performed to detect potential fructose intolerance

Exclusion Criteria:

* smoking,
* fructose intolerance/ -malabsorption,
* pregnancy
* chronic gastrointestinal diseases (e.g. chronic inflammatory bowel disease, irritable bowel syndrome, celiac disease etc.),
* operation on the gastrointestinal tract (exclusively appendectomy)
* anemia,
* hepatic or renal disease
* diabetes mellitus
* consuming illnesses (e.g. cancer, acquired immunodeficiency syndrome (AIDS)) - drug intake affecting lipid or glucose metabolism (cholesterol- or glucose reducing or antihypertensive drugs, steroids, L-Thyroxin, antidepressants, weight reducing drugs).

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08-15 (Actual); Primary Completion 2009-10-15 (Actual); Study Completion 2009-10-15 (Actual)

PRIMARY OUTCOMES:
metabolite concentration | Participants will be followed for the time of four weeks.
  The primary endpoint is the change of metabolite concentration after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.

SECONDARY OUTCOMES:
fatty liver index | Participants will be followed for the time of four weeks.
  Change in fatty liver index after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
Non-alcoholic fatty liver disease (NAFLD) | Participants will be followed for the time of four weeks.
  Change in the classification of non-alcoholic fatty liver disease (NAFLD) based on ultrasound after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
Body weight | Participants will be followed for the time of four weeks.
  Change from baseline in body weight after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
Blood pressure (systolic and diastolic) | Participants will be followed for the time of four weeks.
  Change in blood pressure (systolic and diastolic) after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
GGT | Participants will be followed for the time of four weeks.
  Change in GGT after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
GOT | Participants will be followed for the time of four weeks.
  Change in GOT after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
GPT | Participants will be followed for the time of four weeks.
  Change in GPT after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
AP | Participants will be followed for the time of four weeks.
  Change in AP after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
Triglycerides | Participants will be followed for the time of four weeks.
  Change in triglycerides after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
HDL | Participants will be followed for the time of four weeks.
  Change in HDL after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
LDL | Participants will be followed for the time of four weeks.
  Change in LDL after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
Fasting glucose | Participants will be followed for the time of four weeks.
  Change in fasting glucose after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
BSR | Participants will be followed for the time of four weeks.
  Change in BSR after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
Kreatinine | Participants will be followed for the time of four weeks.
  Change in Kreatinine after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
Uric acid | Participants will be followed for the time of four weeks.
  Change in uric acid after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
Urea | Participants will be followed for the time of four weeks.
  Change in urea after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
Cholesterol | Participants will be followed for the time of four weeks.
  Change in cholesterol after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
Ghrelin | Participants will be followed for the time of four weeks.
  Change in ghrelin after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.
Leptin | Participants will be followed for the time of four weeks.
  Change in leptin after low fructose diet week 1, fruit rich diet, low fructose diet week 3 and HFCS rich diet.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C Bischoff, Principal Investigator — University of Hohenheim

IPD SHARING:
Plan to Share IPD: Undecided